CLINICAL TRIAL: NCT06188286
Title: Patient-Controlled Transcutaneous Acupoint Electrical Stimulation to Improve Quality of Life in Patients With Cancer Pain
Brief Title: The Effect of Patient-Controlled TEAS vs Sham TEAS for Improve Quality of Life in Patients With Cancer Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Liang (Other)
Responsible Party: Sponsor-Investigator, Yi Liang, Principal Investigator, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0593
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Cancer Pain
Keywords: transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS (Active Comparator): transcutaneous acupoint electrical stimulation was performed at the bilateral Hegu and Waiguan acupoints for 30 minutes, and then transcutaneous acupoint electrical stimulation was performed at the Sanyinjiao and Zusanli acupoints of the bilateral lower limbs for 30 minutes.
  Interventions: Other: Transcutaneous electrical acupoint stimulation
- sham TEAS (Placebo Comparator): Except for the transcutaneous acupoint electrical stimulator, which has no current output, the other operations are the same as TEAS group
  Interventions: Other: sham Transcutaneous electrical acupoint stimulation

INTERVENTIONS:
Other: Transcutaneous electrical acupoint stimulation — The 4 patches of the transcutaneous acupoint electrical stimulator were pasted on two pairs of acupuncture points, the output frequency was adjusted to 2Hz, the intensity was up to 50ma, the single intervention time was 30 minutes, and another group of acupuncture points was replaced after completion, and the rest of the operations were the same as above, with a total intervention time of 1 hour.
  Arms: TEAS
Other: sham Transcutaneous electrical acupoint stimulation — The patch is fixed on the acupuncture point to turn on the instrument, but there is no current output
  Arms: sham TEAS

SUMMARY:
The conduct of a pilot trial is of great significance as a means of assessing the feasibility and harmonization of the research and is a very necessary precursor to the better conduct of formal trials. The primary aim of this pilot study is to assess the feasibility of a PC-TEAS in improving the quality of life of cancer patients with pain, with the aspiration of providing process evidence base and an assessment of the intervention for conducting a formal trial. the secondary outcome is to assess the clinical efficacy of the PC-TEAS.

ELIGIBILITY:
Participants who had been diagnosed with cancer pain were eligible if they ①were 18 to 75 years old, ②had NRS pain score of ≥4 in the previous 1 week, or had regular use of analgesics, ③ anticipated survival of at least 6 months, ④ECOG-PS score ≤2 points, ⑤stable vital signs, clear consciousness, and the ability to correctly judge their pain, communication is unhindered, able to cooperate with researchers to complete relevant research assessments, ⑥voluntarily participate in this study and sign the informed consent form. Exclusion criteria included the following: ①Have venous thrombosis of the upper and lower limbs (below the elbow/knee joint), active cerebrovascular disease, severe cardiopulmonary dysfunction, or patient is clinically unstable (eg, acute infections, electrolyte disturbances).②Patients with pacemaker implantation or metal implantation in the body. ③People with local skin at acupoints lesions, poor skin conditions, or other people unsuitable for PC-TEAS treatment. ④Cancer patients who are planning to become pregnant recently or are pregnant. ⑤Have a psychiatric disorder or severe cognitive impairment who are unable to communicate. ⑥Participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Trial feasibility | week 4
  The feasibility of the proposed approach will be evaluated by the number who agreed to participate in the trial.

SECONDARY OUTCOMES:
the changes of EORTC QLQ-C30 score from baseline | week 4, week 8, week 12
  EORTC QLQ-C30 is a specific scale for the quality of life of cancer patients and contains 30 questions. It encompasses three dimensions of assessment which are global quality of life assessment, function assessment (physical, role, emotional, cognitive, social), and symptom assessment (fatigue, nausea, vomiting, pain, dyspnea, sleep, appetite, constipation, diarrhea, and financial). Standardized scores with values ranging from 0 to 100. Higher scores in global quality of life and functioning are indicative of an improved quality of life, whereas higher scores in symptom are associated with poorer health outcomes.
the changes in BPI score of mean pain, severe Pain, least pain and current pain from baesline | week 4, week 8, week 12
  Brief Pain Inventory (BPI) scale is a commonly used scale for evaluating pain. Assess the patient's mean pain, severe pain, least pain score over the past week, and current level of pain. Scores range from 1-10, with higher scores indicating more severe pain.
the amounts of analgesics used | week 4, week 8, week 12
  Changes in Patient Medication Dosage Compared to Baseline.
Index of spontaneous bowel movements | week 4, week 8, week 12
  Spontaneous bowel movements (SBM) refer to bowel movements that have occurred within the past 24 hours without the use of laxatives.Record the number of spontaneous bowel movements of the subject in the past week. Bowel Function Index (BFI) in clinical practice. Specially used to evaluate constipation caused by opioid drugs, the subject's difficulty in defecation and feeling of incomplete defecation in the past week will be recorded. The overall satisfaction rating of defecation.
The changes in mood scale scores of Hamilton Rating Scale for Depression (HAM-D) | week 4, week 8, week 12
  HAM-D is a standardized scale for the measurement of the severity of depressive symptoms, initially designed to yield a total score based on 17 items. The scores of anxiety/depression and its change during the previous 2 weeks from baseline will be recorded.The total score > 24 points, severe depression. 17≤ score ≤24, moderate depression. 7≤ score ≤17, mild depression. < 7 points, no depressive symptoms.
The changes in mood scale scores of Hamilton Rating Scale for Hamilton Rating Scale for Anxiety (HAM-A) | week 4, week 8, week 12
  HAM-A is one of the most widely used rating scales to measure the severity of perceived anxiety symptoms. A total of 14 items were included 14 items. The total score ≥29 points, may be severe anxiety. ≥21 points, there must be obvious anxiety. ≥14 points, must have anxiety. ≥7 points, may have anxiety. < 7 points, no anxiety symptoms.

IPD SHARING:
Plan to Share IPD: No